CLINICAL TRIAL: NCT02093806
Title: Clinical Applications of Round Window High Resolution Computerised Tomography Anatomy in Cochlear Implant Surgery
Brief Title: Clinical Applications of Round Window Imaging Anatomy in Cochlear Implant Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MICHAL.LUNTZ, Prof. Michal Luntz, Bnai Zion Medical Center
Other Study IDs: 0140-13-BNZ; 0140-13-BNZ (Other Grant/Funding Number: TRADIS GAT LTD. ISRAEL)
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Sensorineural Hearing Loss (Disorder)
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CT of the temporal bone
  Interventions: Other: measurment

INTERVENTIONS:
Other: measurment

SUMMARY:
The purpose of this study is to measure the size of the round window niche and its relation to the mastoid segment of the facial nerve and the mastoid cortex, using high resolution computerized tomography of the temporal bone, in order to assess preoperatively what is the extent of obstruction of the round window membrane and whether there is a surgical possibility of round window approach in the insertion of electrode array into the cochlea

DETAILED DESCRIPTION:
The assessment of the anatomy of the round window will be executed using the stractured measuring software used for imaging of the Bnai Zion medical center (CARESTREAM PACS Ver. 11.0, CARSTREAM HEALTH INC.) in IAC window (centered at 700 with a total width of 4000) in the available zoom by the software (usually 400-800%).

Measuring the length (mm) and angle will be executed by the software's structured rulers.

Measuring protocol:

1. Measured scans: one taken in an orbito-meatal plane
2. Chosen slices: where both the round window niche and the external ear canal are seen on the same slice
3. Distances measured:

   1. Distance 1: between the anterior edge of the round window niche and the cortex of the mastoid, with a minimal distance of 0.5mm to the posterior wall of the external ear canal
   2. Distance 2: between the posterior edge of the round window niche and the cortex of the mastoid, with a minimal distance of 0.3mm to the anterior edge of the mastoid segment of the facial nerve.
   3. Distance 3: the size of the round window niche (from its anterior to posterior edges)
   4. Distance 4: between the anterior (most medial) edge of the round window membrane to a point at least 0.3mm anterior to the mastoid segment of the facial nerve.
   5. Distance 5: between the posterior (most lateral) edge of the round window membrane to a point at least 0.3mm anterior to the mastoid segment of the facial nerve
   6. Distance 6: size of round window membrane (anterior/medial to posterior/lateral)
   7. Distance 7: between the lateral edges of distance 1 and 2 marking the cortical size of the "working channel" created between the lines (from the cortex to the round window).
4. Angles measured:

   1. Between distance 1 and 7 - marking the angle of the "working channel" relatively to the cortex
   2. Between distance 1, passing in the middle of distance 3 to the middle of distance 6 - marking the angle of possible insertion from the working channel into the cochlea

ELIGIBILITY:
Inclusion Criteria:

* age 20 years old or older
* high resolution computerized tomography of the temporal bone (slices ≤1mm) before the surgery
* on the measured slices both the round window niche and the posterior wall of the external ear canal are seen

Exclusion Criteria:

* inner, middle or external ear malformation
* temporal bone malformation
* status post cochlear implant
* status post temporal bone trauma
* slices were the round window niche and the posterior wall of the external ear canal are not seen on the same slice

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patient who were suffering from profound sensory neural hearing loss and underwent a high resolution computerized tomography of the temporal bone prior to cochlear implantation surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the size of round window niche and its relation to the cochlea | january-june 2014 (six months)

SECONDARY OUTCOMES:
sizes of working channel from the mastoid cortex into the round window membrane and its relation to the mastoid sagment of the facial nerve | january-june 2014 (six months)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Luntz, Prof., Principal Investigator — chair of otorhinolaryngology department at the Bnai Zion medical center
Locations (1):
- Bnai Zion medical center, Haifa, Israel